CLINICAL TRIAL: NCT01602900
Title: An Open Label Positron Emission Tomography Study in Healthy Male Subjects to Investigate Brain PDE4 Engagement, Pharmacokinetics and Safety of Single Oral Doses of GSK356278, Using 11C-(R)-Rolipram as a PET Ligand(s)
Brief Title: Healthy Volunteer Positron Emission Tomography (PET) Brain Occupancy Study of a Phosphodiesterase 4 (PDE4) Inhibitor in Huntington's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116038
Record Dates: First submitted 2011-12-01; First posted 2012-05-21 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — 5-(5-((2,4-dimethylthiazol-5-yl)methyl)-1,3,4-oxadiazol-2-yl)-1-ethyl-N-(tetrahydro-2H-pyran-4-yl)-1H-pyrazolo(3,4-b)pyridin-4-amine; Rolipram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK356278 (Experimental): Investigational drug
  Interventions: Drug: GSK356278; Drug: Rolipram

INTERVENTIONS:
Drug: GSK356278 — Investigational Medicinal Product
Drug: Rolipram — Challenge Agent

SUMMARY:
This study will investigate if a new experimental drug to treat Huntington's Disease gets into the brain. If it does get into the brain the study will explore the relationship between the amount of drug in the brain and the amount of drug in the blood. The study will involve healthy male volunteers.

DETAILED DESCRIPTION:
This is an open label, non-randomized, adaptive design PET occupancy study in healthy adult males. The primary aim of this study is to describe the relationship between plasma concentrations and brain PDE4 occupancy of GSK356278 over time. Up to 24 healthy volunteers may be administered single doses of GSK356278 in order to obtain 12 evaluable complete data sets of occupancy estimates. This study will help to optimize the dose selection for future clinical studies with GSK356278.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, aged 22-55 years.
* Normal blood pressure, laboratory values, and body mass index
* Willing to agree to study procedures & contraception requirements
* Capable of giving written informed consent

Exclusion Criteria:

* Any evidence of disease that would preclude participation in the clinical study (includes sexually transmitted diseases, exessive alcohol consumption, and substance abuse).
* Previously involved in another clinical trial within 3 months prior to scheduled administration of study drug
* Smoker
* Suffers from claustrophobia
* Any contraindications for MRI scanning (e.g. pacemaker, metal implants or fillings)

Ages: 22 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2012-04-12 (Actual); Study Completion 2012-04-12 (Actual)

PRIMARY OUTCOMES:
Positron Gamma-ray emmision & voxel counts | 60 minutes
  Brain regions of interest and associated radionuclitide-activity
systemic plasma concentration | 24 hours
  serial sampling: GSK356278 concentration expressed as mass per unit of volume

SECONDARY OUTCOMES:
Blood pressure - mm/Hg | 24 hours
  Standard clinical pharmacology safety monitoring of vital signs
ECG - 12-Lead & Telemetry | 24 & 72 hours
  Standard clinical pharmacology safety monitoring
Heart rate - bpm | 72 hours
  Standard clinical pharmacology safety monitoring of vital signs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116038 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116038?search=study&search_terms=116038#rs
- Available data/document: Annotated Case Report Form: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116038 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register